CLINICAL TRIAL: NCT05707156
Title: Prospective Observational Study on the Incidence of Opportunistic Fungal Infections Among Non-HIV Non Transplant Patients by Systemic Corticosteroids Dose
Brief Title: Prospective Observational Study on the Incidence of Opportunistic Fungal Infections
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Georgia (Other); University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 18-2577
Record Dates: First submitted 2023-01-20; First posted 2023-01-31 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Pneumocystis Jirovecii Infection; Pneumocystis; Cryptococcosis; Candidiasis; Aspergillosis
Keywords: Immunocompetent; Corticosteroids; Pneumocystis carinii; Pneumocystis jirovecii; mortality; HIV-negative patients
MeSH Terms: conditions — Pneumocystis Infections; Pneumonia, Pneumocystis; Cryptococcosis; Candidiasis; Aspergillosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Low dose: Cumulative dose of corticosteroids 0-10 mg a day (prednisone equivalent) Prednisone: 0-10 mg OR, Dexamethasone: 0-1.5 mg OR, Prednisolone: 0-10 mg OR, Methylprednisolone: 0-8 mg
- Medium dose: Cumulative dose of corticosteroids 10-20 mg a day (prednisone equivalent):
  Prednisone: 11-20 mg OR, Dexamethasone: 1.6-3.0 mg OR, Prednisolone: 11-20 mg OR, Methylprednisolone: 9-16 mg
- High dose: Cumulative dose of corticosteroid >20 mg a day (prednisone equivalent):
  Prednisone: > 20 mg OR, Dexamethasone: > 3.0 mg OR, Prednisolone: > 20 mg OR, Methylprednisolone: >16 mg

SUMMARY:
Corticosteroids exposure is a common risk factor for invasive fungal infections. Systemic corticosteroid therapy treats several medical conditions, including rejection in solid organ transplant recipients, malignancy, and autoimmune or inflammatory diseases. Corticosteroid exposure is a well-known risk factor for developing PJP. Still, it remains unclear how prior corticosteroid exposure influences the presentation, severity, and mortality of opportunistic fungal infections. The investigators aim to prospectively characterize the corticosteroid use as a dose response to inform risk of invasive fungal infections.

DETAILED DESCRIPTION:
The investigators will use TriNetX, a global federated research network that captures anonymous data from electronic medical records (EMRs) of 66 healthcare organizations. The investigators are setting up a prospective observation study of non-HIV, non-transplant (NHNT) patients who are receiving systemic (oral or intravenous) corticosteroids for more than 2 weeks. The investigators are planning on excluding individuals younger than 18 years old with any prior history of Cryptococcosis, Aspergillosis, Pneumocystis jirovecii pneumonia or invasive candidiasis. The investigators will follow 3 cohorts of patients based on their daily cumulative prednisone equivalent dose in mg. Group 1: 0-10 mg a day, group 2: 10-20 mg a day, group 3: > 20 mg daily. The investigators will record any incidence of Cryptococcosis, Aspergillosis, Pneumocystis jirovecii pneumonia or invasive candidiasis based on ICD-10 codes or labs results at 3-6 months intervals. The investigators will record as well additional clinical features for patients including demographics, comorbidities, medications, and limited labs.

ELIGIBILITY:
Inclusion Criteria:

* Patients on systemic corticosteroids for more than 2 weeks

Exclusion Criteria:

* HIV infection
* Transplant status
* Younger than 18 years of age
* Previous history of Cryptococcosis, Aspergillosis, Pneumocystis jirovecii pneumonia or invasive candidiasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-HIV, non-transplant immunocompromised individuals on systemic corticosteroids
Sampling Method: Non-Probability Sample
Enrollment: 12032 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
PJP | 3-6 months after first corticosteroid use
  Number of cases of Pneumocystis jirovecii pneumonia
Cryptococcosis | 3-6 months after first corticosteroid use
  Number of cases of cryptococcosis
Aspergillosis | 3-6 months after first corticosteroid use
  Number of cases of Aspergillosis
Candidiasis | 3-6 months after first corticosteroid use
  Number of cases of Candidiasis

SECONDARY OUTCOMES:
Mortality | 3-6 months after first corticosteroid use
  Number of deaths
Hospitalization | 3-6 months after first corticosteroid use
  Number of hospitalization episodes

CONTACTS AND LOCATIONS:
Overall Officials: ANDRES F HENAO, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- TrinetX based global network, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Not available, not applicable

REFERENCES:
- [Result] Mundo W, Morales-Shnaider L, Tewahade S, Wagner E, Archuleta S, Bandali M, Chadalawada S, Johnson SC, Franco-Paredes C, Shapiro L, Henao-Martinez AF. Lower Mortality Associated With Adjuvant Corticosteroid Therapy in Non-HIV-Infected Patients With Pneumocystis jirovecii Pneumonia: A Single-Institution Retrospective US Cohort Study. Open Forum Infect Dis. 2020 Aug 13;7(9):ofaa354. doi: 10.1093/ofid/ofaa354. eCollection 2020 Sep. PMID 33005696
- [Result] Gharamti AA, Mundo W, Chastain DB, Franco-Paredes C, Henao-Martinez AF, Shapiro L. Pneumocystis jirovecii pneumonia: a proposed novel model of corticosteroid benefit. Ther Adv Infect Dis. 2021 Jul 20;8:20499361211032034. doi: 10.1177/20499361211032034. eCollection 2021 Jan-Dec. No abstract available. PMID 34349985
- [Result] Chastain DB, Kung VM, Golpayegany S, Jackson BT, Franco-Paredes C, Vargas Barahona L, Thompson GR 3rd, Henao-Martinez AF. Cryptococcosis among hospitalised patients with COVID-19: A multicentre research network study. Mycoses. 2022 Aug;65(8):815-823. doi: 10.1111/myc.13476. Epub 2022 Jun 19. PMID 35657109